CLINICAL TRIAL: NCT01632644
Title: Pilot Study of Skin Biopsy Sites: A Consensus Approach Based on Patient and Physician Interviews
Brief Title: Identifying Skin Biopsy Sites
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Other Study IDs: STU66384
Record Dates: First submitted 2012-06-27; First posted 2012-07-03 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Identification of Skin Cancer Biopsy Sites
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Physicians: Physicians performing skin biopsies
  Interventions: Other: Survey/Interview
- Patients: Patients who have had skin biopsies
  Interventions: Other: Survey/Interview

INTERVENTIONS:
Other: Survey/Interview — Each group will be surveyed and interviewed.

SUMMARY:
The primary objective of this study is to investigate the patient experience during skin biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and Over
* The subjects are in good health.
* The subjects have the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.
* Patients who have had one or multiple skin biopsies OR board-certified dermatologists.

Exclusion Criteria:

* Under 18 years of age.
* Subjects who are unable to understand the protocol or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians will be recruited by email obtained through directories.
  Patients will be those who have had biopsies at the Northwestern University Department of Dermatology.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Review of Physician and Patient Experience | Last four weeks of study
  Subjects will answer a combination of:
  1. Open-ended questions and
  2. Questions asking for subject to rank possible responses

SECONDARY OUTCOMES:
Physician's Experience with Skin Biopsy Sites | First four weeks of study
  Physicians will answer a combination of:
  1. Open-ended questions, and
  2. Questions asking for subject to rank possible responses
Patient's Experience with Skin Biopsy Sites | First four weeks of study
  Patients will answer a combination of:
  1. Open-ended questions and
  2. Questions asking for subject to rank possible responses

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Dermatology, Chicago, Illinois, United States